CLINICAL TRIAL: NCT02592161
Title: A Randomized, Single Center, Double Blind, Parallel, Placebo-controlled Clinical Study of Efficacy and Safety of Chung A Won in Women's Patients With Osteoporosis
Brief Title: Clinical Study of Efficacy and Safety of Chung A Won in Women's Patients With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Hyun Lee, Professor, Korea Health Industry Development Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B110051; NCT01771510 (obsolete NCT alias)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Test drug : Granules, Chung A Won 3g (Eucommiaceae, Psoralea corylifolia, Walnut, Ginger) Three times a day, oral administration for 24weeks
  Interventions: Drug: Experimental
- Placebo comparator (Placebo Comparator): Reference drug : Granules, Placebo 3g (Lactose hydrate, Corn starch, Caramel pigment) Three times a day, oral administration for 24weeks
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Experimental — Test drug : Granules, Chung A Won 3g (Eucommiaceae, Psoralea corylifolia, Walnut, Ginger) Three times a day, oral administration for 24weeks
  Reference drug : Granules, Placebo 3g (Lactose hydrate, Corn starch, Caramel pigment)
  Three times a day, oral administration for 24weeks
  Other Names: Chung A Won

SUMMARY:
A randomized, single center, double blind, parallel, placebo-controlled, clinical study of efficacy and safety of Chung A Won and placebo for 24 weeks three times a day on the improvement of osteoporosis and symptoms in Women's older than 50 patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1)Female more than 50 years old in osteoporosis

Exclusion Criteria:

1. Wash out peroid: using agents more than 3 months against osteoporosis
2. Subject who takes drugs that may affect the clinical trials (Corticosteroids, anticonvulsants, tranquilizers, antidepressants, hypnotic, diuretic)
3. Subject who has a chronic liver disease, thyroid disease and chronic renal disease
4. Subject who is chronic alcoholics and undernourished
5. Other conditions were not suitable in study : Severe physical defects mental defects
6. Pregnant woman
7. Subject who is not calibrated hypercalcemia/hypocalcemia
8. Secondary osteoporosis : Subject who takes drugs(Glucocorticoid, Diabetes Medications)
9. Subject who has 60% more fracture risk in FRAX(WHO fracture risk assessment tool)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The change of T-score of bone mineral density(QCT) | baseline, After 24 weeks(± 3 days) from the baseline of the trial

SECONDARY OUTCOMES:
The change of T-score | baseline, After 4 weeks, 12 weeks from the baseline of the trial
The change of osteoporosis-related indicators of blood tests | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial
The change of ODI(Oswestry Disability Index) | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial
The change of QVAS(Quardruple Visual Analog Scale) | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial
The change of kupperman index | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial
The change of shin-huh symptoms | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial
The change of quality of life using SF-36 | baseline, After 4 weeks, 12 weeks, 24 weeks(endpoint) from the baseline of the trial